CLINICAL TRIAL: NCT03984968
Title: Evaluation of the Safety and Efficacy of CD19 CAR-T Combined With Autologous T Cells Engineered to Express CD19 (CD19+ Feeding T Cells, FTCs) for Consolidation Treatment for Acute Lymphoblastic Leukemia
Brief Title: CD19 CAR-T Consolidation Therapy for Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SZCART01
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia, Adult B-Cell
Keywords: feeding T cell; CD19 CAR-T therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FTCs: High dose (Phase 1) (Experimental)
  Interventions: Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion
- FTCs: Medium dose (Phase 1) (Experimental)
  Interventions: Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion
- FTCs: Low dose (Phase 1) (Experimental)
  Interventions: Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion
- FTCs: High dose (Phase 2) (Experimental)
  Interventions: Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion

INTERVENTIONS:
Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion — Phase 1: Optimal biological doses of feeding T cells (FTCs) identification. ssCART-19 cells combined with CD19+ FTCs were administered to Philadelphia chromosome-positive B-ALL patients with remission. ssCART-19 was infused at the dose of 5×10^6/kg on days 1 to 3 of the first cycle and on day 1 of the second to fourth cycle. CD19+ FTCs (5×10^6 cells/kg) were infused two hours after the infusion of ssCART-19 cells on day 1 and at the same dose alone on day 8 of the second to fourth cycle. Five patients were enrolled in this arm, and all the patients received four cycles of ssCART-19 consolidation.
  Arms: FTCs: High dose (Phase 1)
Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion — Phase 1: Optimal biological doses of feeding T cells (FTCs) identification. ssCART-19 cells combined with CD19+ FTCs were administered to Philadelphia chromosome-positive B-ALL patients with remission. ssCART-19 was infused at the dose of 5×10^6/kg on days 1 to 3 of the first cycle and on day 1 of the second to fourth cycle. CD19+ FTCs (3.25×10^6 cells/kg) were infused two hours after the infusion of ssCART-19 cells on day 1 and at the same dose alone on day 8 of the second to fourth cycle. Four patients were enrolled in this arm, and all the patients received four cycles of ssCART-19 consolidation.
  Arms: FTCs: Medium dose (Phase 1)
Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion — Phase 1: Optimal biological doses of feeding T cells (FTCs) identification. ssCART-19 cells combined with CD19+ FTCs were administered to Philadelphia chromosome-positive B-ALL patients with remission. ssCART-19 was infused at the dose of 5×10^6/kg on days 1 to 3 of the first cycle and on day 1 of the second to fourth cycle. CD19+ FTCs (2×10^6 cells/kg) were infused two hours after the infusion of ssCART-19 cells on day 1 and at the same dose alone on day 8 of the second to fourth cycle. Four patients were enrolled in this arm, and all the patients received four cycles of ssCART-19 consolidation.
  Arms: FTCs: Low dose (Phase 1)
Biological: ssCART-19 cells combined with CD19+ feeding T cells (FTCs) infusion — Phase 2: Expansion Study. ssCART-19 cells combined with FTCs at the optimal biological dosage determined in the Phase 1 study were given to expanded Philadelphia chromosome-positive B-ALL patients with remission. The 5×10^6 cells/kg of CD19+ FTCs was the optimal biological dose determined in phase I. Therefore, CD19+ FTCs at 5×10^6 cells/kg were infused two hours after the infusion of ssCART-19 cells on day 1 and at the same dose alone on day 8 of the second to fourth cycle, while ssCART-19 was infused at the dose of 5×10^6/kg on days 1 to 3 of the first cycle and on day 1 of the second to fourth cycle. The Bayesian optimal design was applied to perform the futility assessment at the specified interim analyses. Thirty-four evaluable subjects were recruited, and all the patients received at least two cycles of ssCART-19 consolidation.
  Arms: FTCs: High dose (Phase 2)

SUMMARY:
This is a single-arm, open-label, single-center, phase I/II study to determine the safety and efficacy of CD19 CAR-T(ssCART-19) combined with autologous T cells engineered to express CD19, namely CD19+ feeding T cells (FTCs), as consolidation therapy in patients diagnosed with de novo Philadelphia chromosome-positive CD19+ B-ALL.

The study will contain the following sequential phases: screening, lymphocyte apheresis, induction, and consolidation chemotherapies combined with tyrosine kinase inhibitors. Once in complete response, patients will receive two to four cycles of ssCART-19s, namely one cycle of ssCART-19 infusion (CAR-T1) followed by one to three cycles of ssCART-19 and CD19+ FTC infusion (CAR-T2-4). The role of CD19+ FTCs is to mimic leukemia cells. Therefore, they are expected to stimulate in vivo expansion and persistence of ssCART-19.

Considering the limited number of lymphocytes obtained by a single apheresis from patients and cost-efficacy, in addition to safety, we will explore the range of biologically active doses of FTCs in a phase I study. Based on preclinical data, FTCs' stimulation of ssCART-19 at a ratio of 1:1 could achieve the best activation response, so a 5×10^6/kg dosage of FTCs was set as the initial dosage in the study, and lower doses were also evaluated. In phase I, FTCs will be administered at the dose of 5×10^6/kg, 3.25×10^6/kg, or 2×10^6/kg two hours after ssCART-19 infusion on day 1 and once again administered at the same dose on day 8. After ssCART-19 and FTCs infusion, adverse events (AEs) as the primary endpoints will be recorded for 6 months; efficacy as the secondary endpoint will be assessed by detecting molecular response for 6 months, PFS, and OS for 2 years.

In phase II, we will expand the study at optimal biological doses of FTCs and further evaluate the efficacy and safety of the innovative combination therapy of ssCART-19 and FTCs. The primary endpoint was the complete molecular response (CMR). The secondary endpoints were RFS, OS, and adverse events (AEs) of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 15-65 years of age at the time of signing informed consent
* Diagnosed as de novo Philadelphia chromosome-positive CD19+ B-ALL
* Karnofsky performance status ≥ 60 or Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Unable to find a suitable donor or for other reasons to undergo allogeneic hematopoietic stem cell transplantation during the study
* Ability and willingness to adhere to the study visit schedule and all protocol requirements
* Voluntarily sign informed consent forms

Exclusion Criteria:

* Unable to tolerate any kind of TKIs (including the first- and second-generation tyrosine kinase inhibitors) for a long period.
* Subjects who have positive mutation(s) of the ABL kinase domain and require the third-generation tyrosine kinase inhibitors for long-term therapies.
* Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 × upper limit of normal (ULN) and direct bilirubin > 1.5 × ULN
* Inadequate renal function defined by serum creatinine > 1.6 mg/dL
* International ratio (INR) or partial thromboplastin time (PTT) > 1.5 x ULN
* Left ventricular ejection fraction < 50%
* Ongoing treatment with chronic immunosuppressants
* Significant comorbid conditions or diseases which, in the judgment of the investigator, would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, recent significant traumatic injury, and other conditions
* Known human immunodeficiency virus (HIV) positivity
* Subjects with a history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control
* Subjects with second malignancies in addition to ALL
* Pregnant or lactating women, or subjects refusing to take effective contraception measures
* Other contraindications that are considered inappropriate to participate in this trial

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2040-01-24 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Incidence of adverse events (AEs) and abnormal laboratory test results | 6 months after ssCART-19 consolidation termination (CAR-T4; each cycle is 3 months)
  AEs will be assessed according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE5.0).
Phase 2 Molecular response after CD19 CAR-T consolidation therapy combined with CD19+ feeding T cells | 3 months after each cycle of ssCART-19 consolidation termination (each cycle is 3 months)
  Complete molecular response (CMR) was defined as the absence of a detectable BCR-ABL1 transcript with a sensitivity of 0.01%.

SECONDARY OUTCOMES:
Phase 1 Molecular response after CD19 CAR-T consolidation therapy combined with CD19+ feeding T cells. | 3 months after each cycle of ssCART-19 consolidation termination (each cycle is 3 months)
  Complete molecular response (CMR) was defined as the absence of a detectable BCR-ABL1 transcript with a sensitivity of 0.01%.
Phase 1 The range of biologically active doses and optimal biological doses of CD19+ feeding T cells. | 6 months after ssCART-19 consolidation termination (CAR-T4; each cycle is 3 months)
  The range of biologically active doses and optimal biological doses of CD19+ feeding T cells will be determined.
Phase 1 Overall survial (OS) | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Phase 1 Relapse free survival（RFS） | 2 years
  It is measured from the date of achievement of a remission until the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.
Phase 2 Incidence of adverse events (AEs) and abnormal laboratory test results | 6 months after ssCART-19 consolidation termination (the specific date depending how many cycles the participants received; each cycle is 3 months)
  AEs will be assessed according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE5.0).
Phase 2 Overall survial (OS) | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Phase 2 Relapse free survival（RFS） | 2 years
  It is measured from the date of achievement of a remission until the date of relapse from CR, or CRi, or death from any cause; patients not known to have any of these events are censored on the date they were last examined.

OTHER OUTCOMES:
Phase 1 exploratory endpoints | 3 months after ssCART-19 consolidation termination (CAR-T4; each cycle is 3 months)
  Assessment of persistence of CD19+ FTCs, and expansion and persistence of ssCART-19 cells in the peripheral blood
Phase 1 exploratory endpoints | Two weeks during each cycle of ssCART-19 (CAR-T1-4; each cycle is 3 months)
  Evaluate cytokine/chemokine induction in the blood of subjects after infusion of CD19+ FTCs and CD19 CAR-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics of patients, outcomes
Supporting Information: SAP, CSR
Time Frame: One year after the study termination
Access Criteria: Clinical researchers worldwide can access the IPD and supporting information after author authorization. They can get IPD details by visiting the ResMan system.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Derived] Chen LY, Gong WJ, Li MH, Zhou HX, Xu MZ, Qian CS, Kang LQ, Xu N, Yu Z, Qiao M, Zhang TT, Zhang L, Tian ZL, Sun AN, Yu L, Wu DP, Xue SL. Anti-CD19 CAR T-cell consolidation therapy combined with CD19+ feeding T cells and TKI for Ph+ acute lymphoblastic leukemia. Blood Adv. 2023 Sep 12;7(17):4913-4925. doi: 10.1182/bloodadvances.2022009072. PMID 36897251